CLINICAL TRIAL: NCT02601404
Title: REal World Advanced Experience of BioResorbable ScaffolD by SMart Angioplasty Research Team (SMART REWARD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, MD,PhD, Samsung Medical Center
Other Study IDs: 2015-07-163
Record Dates: First submitted 2015-11-05; First posted 2015-11-10 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bioresorbable Scaffold: Patients receiving percutaneous coronary intervention (PCI) for coronary artery disease using Absorb™(Abbott Vascular)
  Interventions: Device: Bioresorbable scaffold (BRS)

INTERVENTIONS:
Device: Bioresorbable scaffold (BRS) — The implantation procedure of an Absorb™ is similar to a metallic stent.
  Other Names: Absorb™ (Abbott Vascular)

SUMMARY:
Current drug-eluting stents (DES) has demonstrated excellent clinical outcomes in patients with coronary artery disease. However, a continued risk of clinical events even several years after the procedure is reported. Stent platform or polymer-associated inflammation may play a role.

Bioresorbable scaffold (BRS) is known to disappear 2 to 3 years after the implantation, which may result in the more favorable very long-term clinical outcomes compared with metallic stents. The initial clinical experiences of BRS in relatively simple lesion subsets were comparable to DESs.

BRS, however, is limited by the disadvantageous mechanical characteristics such as thick strut and the risk of fracture by overdilation. There is concern that BRS is less optimal for complex lesion subsets such as bifurcation lesions, calcified tortuous lesions, or diffuse long lesions. Real world registry is needed to test the feasibility and safety of BRS in these complex lesion subsets.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 19 and 70 years old.
* Patients with a significant lesion in a de novo coronary artery: a percent diameter stenosis (DS) 50% with 1) a positive history of recurrent angina pectoris; (2) objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent); or (3) abnormal results of any invasive functional diagnostic test (eg, fractional flow reserve) or a percent DS ≥70% even in the absence of the above-mentioned ischemic signs or symptoms.
* Patients are scheduled for coronary intervention
* He/she or his/her legally authorized representative provides written informed consent

Exclusion Criteria:

* Experience of cardiopulmonary resuscitation
* Cardiogenic shock
* Expected survival less than 2 years
* Pregnancy or breast feeding
* Opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 1,000 patients derived from a population of Korean patients receiving PCI for coronary artery disease will be enrolled in the present registry. It is recommended that each enrolling investigator review the most recent instructions for use (IFU) of Absorb™ and assess the contraindications, warnings, and precaution sections for treating potential patients.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
cardiac death | 2 years
  Target vessel failure (TVF) of cardiac death, myocardial infarction (MI) attributed to the target vessel, and target vessel revascularization (TVR)

SECONDARY OUTCOMES:
Device success | maximum of 7 days
  Successful delivery and deployment of the study scaffold at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold residual stenosis of less than 30% by quantitative coronary angiography (QCA) (by visual estimation if QCA unavailable).
Procedural success | maximum of 7 days
  Achievement of final in-scaffold residual stenosis of less than 30% by QCA (by visual estimation if QCA unavailable) with successful delivery and deployment of at least one study scaffold at the intended target lesion and successful withdrawal of the delivery system for all target lesions without the occurrence of cardiac death, target vessel MI or repeat target lesion revascularization (TLR) during the hospital stay (maximum of 7 days).
Target vessel failure (TVF) | 1, 3, and 5 years
  cardiac death, target vessel MI, or TVR
Each component of Target vessel failure (TVF) | 1, 2, 3 and 5 years
  Cardiac death,Vascular death,Non-cardiovascular death,Myocardial Infarction (MI)
Target lesion failure | 1, 2, 3 and 5 years
  Target lesion failure of cardiac death, MI attributed to the target vessel, and Target Lesion Revascularization(TLR). TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches and the target lesion itself.
Definite or probable stent thrombosis | 1, 2, 3 and 5 years
Periprocedural enzyme elevation | 1, 2, 3 and 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiac and Vascular Center; Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee JM, Joh HS, Choi KH, Hong D, Park TK, Yang JH, Song YB, Choi JH, Choi SH, Jeong JO, Lee JY, Choi YJ, Chae JK, Hur SH, Bae JW, Oh JH, Chun KJ, Kim HJ, Cho BR, Shin D, Lee SH, Hwang D, Lee HJ, Jang HJ, Kim HK, Ha SJ, Shin ES, Doh JH, Hahn JY, Gwon HC; SMART-REWARD Investigators. Safety and Efficacy of Everolimus-Eluting Bioresorbable Vascular Scaffold Versus Second-Generation Drug-Eluting Stents in Real-World Practice. J Korean Med Sci. 2023 Feb 6;38(5):e34. doi: 10.3346/jkms.2023.38.e34. PMID 36747363